CLINICAL TRIAL: NCT02028663
Title: A Double-Blind, Randomized, Dose-finding Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Erosive Esophagitis
Brief Title: Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Erosive Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CJ_APA_201
Record Dates: First submitted 2014-01-05; First posted 2014-01-07 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Erosive Esophagitis; GERD
Keywords: P-CAB; APA(Acid Pump Antagonist)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CJ-12420 Amg (Experimental): 50 volunteers will be administered CJ-12420 Amg
  Interventions: Drug: CJ-12420
- CJ-12420 Bmg (Experimental): 50 volunteers will be administered CJ-12420 Bmg
  Interventions: Drug: CJ-12420
- CJ-12420 Cmg (Experimental): 50 volunteers will be administered CJ-12420 Cmg
  Interventions: Drug: CJ-12420
- Esomeprazole 40mg (Active Comparator): 50 volunteers will be administered Esomeprazole 40mg
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: CJ-12420 — Once daily, Oral administration
  Other Names: Undecided
  Arms: CJ-12420 Amg; CJ-12420 Bmg; CJ-12420 Cmg
Drug: Esomeprazole — Once daily, Oral administration
  Other Names: Nexium
  Arms: Esomeprazole 40mg

SUMMARY:
The purpose of this study is to investigate the optimal dose and administration methods of CJ-12420 in patients with erosive esophagitis by comparing the safety and efficacy of orally administered CJ-12420 to esomeprazole 40mg.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-70
* Diagnosed with Erosive Esophagitis by Esophagogastroduodenoscopy (EGD) and classified into LA Grade A to D within 14 days before randomization to treatment

Exclusion Criteria:

* Patients who cannot undergo EGD
* Patients diagnosed with irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), or suspected IBS
* Patients who took PPIs within 2 weeks prior to study drug administration
* Long-term use of nonsteroidal anti-inﬂammatory drugs throughout the study
* Clinically significant abnormal laboratory values during screening

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cumulative healing rate of erosive esophagitis at 8-week | 8 week

SECONDARY OUTCOMES:
Healing rate of erosive esophagitis at 4-week | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Chae Jung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital and 11 others, Seoul, South Korea